CLINICAL TRIAL: NCT06165679
Title: Comparison Between the Effect of Prilocaine vs Bupivacaine on Hemodynamics in Spinal Anesthesia for Geriatric Patients Undergoing Endoscopic Urological Surgeries: A Randomized Controlled Trial
Brief Title: Effect of Prilocaine vs Bupivacaine on Hemodynamics in Spinal Anesthesia for Geriatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdElKhalik Mahmoud Shaban, Lecturer of anaesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N-439-2023
Record Dates: First submitted 2023-12-02; First posted 2023-12-11 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Hemodynamic Instability
MeSH Terms: interventions — Prilocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prilocaine group (Active Comparator)
  Interventions: Drug: Prilocaine
- Bupivacaine GROUP (Active Comparator)
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Prilocaine — The patients will receive a single injection of spinal anesthesia using prilocaine plus fentanyl
  Arms: Prilocaine group
Drug: Bupivacaine — The patients will receive a single injection of spinal anesthesia using Bupivacaine plus fentanyl
  Arms: Bupivacaine GROUP

SUMMARY:
Data comparing prilocaine vs bupivacaine in equipotent doses in the elderly are lacking; therefore, the study will compare the effect of prilocaine vs bupivacaine on hemodynamics in spinal anesthesia for geriatric patients undergoing endoscopic urological surgeries

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years old and above.
* Both genders.
* Patients scheduled to undergo endoscopic urological surgeries.
* ASA I and II class.

Exclusion Criteria:

* Patient refusal.
* Known local anesthetic (LA) allergy.
* Bleeding disorders.
* Skin lesions or infections at site of needle insertion.
* Hypertensive patients.
* Patients candidate for transurethral resection of the prostate
* ASA III and VI class

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Hypotension | Till 30 minutes after spinal anesthesia.
  Incidence of hypotension from local anesthetic injection

SECONDARY OUTCOMES:
Use of vasopressor drugs | Until the patient will have no lower limbs motor weakness assessed up to 6 hours after spinal anesthesia
  Total doses of vasopressor drugs used for hypotension treatment

OTHER OUTCOMES:
Mean and systolic arterial blood pressure values | Until the patient will have no lower limbs motor weakness assessed up to 6 hours after spinal anesthesia
  Mean and systolic arterial blood pressure values after spinal anesthesia
Heart rate | Until the patient will have no lower limbs motor weakness assessed up to 6 hours after spinal anesthesia
  Heart rate after spinal anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini hospital, Cairo, Egypt